CLINICAL TRIAL: NCT03835325
Title: A Multicenter, Non-comparative, Phase IV Clinical Trial Evaluation of the Effect of Cogmax® in the Treatment of Memory Loss in Postmenopausal Women
Brief Title: The Effect of a Multivitamin in the Treatment of Memory Loss in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EF152
Record Dates: First submitted 2018-12-21; First posted 2019-02-08 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Memory Disorders; Postmenopausal Symptoms
Keywords: Postmenopausal Symptoms, Memory Disorders
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cogmax® (Experimental): Research participants will receive 2 capsules of Cogmax® per day (after lunch) for 12 weeks.
  Interventions: Dietary Supplement: Cogmax®

INTERVENTIONS:
Dietary Supplement: Cogmax® — Research participants will receive 2 capsules of Cogmax® per day (after lunch) for 12 weeks.

SUMMARY:
Complaints about memory loss are very common in women in the menopausal transition period. The effectiveness of estrogen replacement therapy in cognitive improvement is controversial. Partial positive results were obtained in some studies with regard to memory improvement, so far no standard treatment considered effective in these cases. Effective pharmacological approaches to the treatment of memory loss associated with menopause are an unmet medical need. Cogmax® is a multivitamin and mineral supplement that contains numerous key elements for cognitive function, and may be a safe therapeutic option in these cases.

The multicenter, non-comparative (single-arm) phase IV clinical trial will be conducted with 80 female participants aged 45 to 60 years and menopausal memory loss complaint.

After 3 months of using multivitamin and mineral supplement, memory and attention will be reevaluated through specific questionnaire and the Stroop Test Victoria version.

DETAILED DESCRIPTION:
This multicenter, non-comparative phase IV clinical trial will be conducted at brazilian clinical trial centers under the auspices of Eurofarma Laboratories S.A. Recruitment for the study will begin after the relevant ethical and regulatory approvals and will have an estimated duration of 4 months.

The study will include 80 female participants aged between 45 and 60 years and menopausal memory complaints who consent to participate in the study by signing the informed consent form.

To be included, participants must meet all inclusion criteria and none of the exclusion criteria. Each participant will initially complete a selection period with a maximum duration of 14 days for evaluation of eligibility. Participants will then be treated with Cogmax® in the dosage of two capsules per day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 45 years and ≤ 60 years.
2. Memory loss associated with menopause.
3. Score ≤ 3.0 (mean value found in the elderly) related to the self-efficacy factor, consisting of the sum of the scores for the Capability, Control and Change domains obtained through the Metamemory in Adulthood Questionnaire - reduced version (MIAr).
4. Amenorrhea for at least 1 year and there is no more than 6 years.
5. Serum FSH dosage> 30mIU / mL.
6. Dosage of serum estradiol <20pg / mL.
7. Knowledge of the Portuguese language sufficient to answer the questionnaires.
8. Signature of the Free and Informed Consent Form (EHIC) prior to any study procedure.

Exclusion criteria:

Individuals who meet at least one of the following criteria will be excluded from the study:

1. Complaints of hot flashes, insomnia and / or very intense sleep disorders, at the discretion of the investigator.
2. Presence of moderate to severe depression, score ≥ 18 at assessment through the Beck Depression Inventory. ,
3. Presence of moderate to severe anxiety, with a ≥ 30 score on the Beck anxiety inventory. ,
4. Initiation of hormone replacement therapy in the 6 months prior to study inclusion. Patients receiving hormone replacement therapy starting more than 6 months before inclusion in the study may be included in the study provided that the treatment is regular with the same drug and the same dose during the last 6 months before inclusion and provided that this treatment is maintained throughout the study.
5. Use of psychotropic medications (anticonvulsants, benzodiazepines, antipsychotics), selective serotonin reuptake inhibitors (SSRIs) and selective serotonin and noradrenaline reuptake inhibitors (SSRIs)
6. Alcoholism and / or use of other illicit drugs.
7. History of allergy or intolerance to any component of the experimental product formulation.
8. Diagnosis of neurological diseases associated with cognitive deficits (including dementia and mental retardation) or psychiatric illnesses.
9. Presence of serious or uncontrolled diseases (such as decompensated hypothyroidism) at the discretion of the researcher (such as stroke, Parkinson's disease, etc.).
10. Participation in clinical research protocol in the previous 12 months unless, at the discretion of the researcher, their participation in the study may incur direct benefit to the research participant.
11. Presence of any condition that, at the discretion of the researcher, makes the patient unfit to participate in the study.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cassiano O Berto, Principal Investigator — Eurofarma Laboratorios S.A.
Locations (1):
- CEPIC, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Beginning of the study: 01/28/2019 (first visit of the first participant) End of study: 12/09/2019 (last visit of the last participant)
  Recruitment´s type of location: Medical clinic
Pre-assignment Details: Inclusion criteria, exclusion criteria and other reasons
Groups:
- Cogmax®: Research participants will receive 2 capsules of Cogmax® per day (after lunch) for 12 weeks.
  Cogmax®: Research participants received 2 capsules of Cogmax® per day (after lunch) for 12 weeks.
Period: Overall Study
Arm/Group | Cogmax®
Started (80 participants aged between 45 and 60 years old and complaining of memory loss associated with menopause.) | 80
Completed | 78
Not Completed | 2
Not completed — Lack of adherence to protocol procedures | 1
Not completed — Selection failure | 1

BASELINE CHARACTERISTICS:
Population: Efficacy analyzes were performed for the population with modified treatment intent (mITT, n=78)
Groups:
- Cogmax®: Cogmax®: Research participants received 2 capsules of Cogmax® per day (after lunch) for 12 weeks.
Arm/Group | Cogmax®
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 80
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 53
  More than one race | 0
  Unknown or Not Reported | 0
Vital signs [Mean (Standard Deviation); unit: mmHg]
  Systolic arterial pressure | 125.0 (15.1)
  Diastolic arterial pressure | 77.4 (10.0)
Heart rate [Mean (Standard Deviation); unit: bpm] | 69.2 (10.6)
respiratory rate [Mean (Standard Deviation); unit: breaths per minute] | 16.6 (1.4)
SELF-EFFICACY Factor [Mean (Standard Deviation); unit: Score] — The baseline measure will evaluate the score relative to the self-efficacy factor (SEF), consisting of arithmetic average on the domains capacity, control and change of the Meta-memory in Adulthood Questionnaire - Portuguese reduced version (MIAr)
  The arithmetic average on the domains capacity, control and change range from 1 (worse) to 5 (better). Population: Efficacy analyzes were performed for the population with modified treatment intent (mITT, n=78)
  Score
    mITT population: number analyzed (Participants) | 78
    mITT population | 2.5 (0.3)
    PP population | 2.5 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of the Score Number Relative to the Self-efficacy Factor, Consisting of Average Scores on the Domains Capacity, Control and Change of the Meta-memory in Adulthood Questionnaire - Portuguese Reduced Version
Description: The primary outcome measure will evaluate the change from baseline in the score relative to the self-efficacy factor (SEF), consisting of arithmetic average on the domains capacity, control and change of the Meta-memory in Adulthood Questionnaire - Portuguese reduced version (MIAr) SEF final - SEF baseline ≤ 0 (no improvement in the measured memory capacity between the initial and final evaluations) SEF final - SEF baseline > 0 (improvement in the memory capacity measured between the initial and final evaluations)
  The arithmetic average on the domains capacity, control and change range from 1 (worse) to 5 (better).
Time Frame: 12 weeks after the start of the treatment (Baseline)
Population: mITT and PP. Efficacy analyzes were performed for the population with modified treatment intent (mITT, n=78)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cogmax®
Number analyzed (Participants) | 80
score on a scale
  mITT: number analyzed (Participants) | 78
  mITT | 2.9 (0.5)
  PP | 2.9 (0.5)
Statistical Analysis 1: Comparison: Cogmax®; The sample size calculation was based on the following hypothesis test: H0: there is no improvement in memory capacity between the initial (VS) and final (VF) assessments, assessed by the self-efficacy factor of the MIAr questionnaire. H1: there is an improvement in memory capacity between the initial (VS) and final (VF) assessments, assessed by the self-efficacy factor of the MIAr questionnaire. or H0: AUTO-EF (VF) - AUTO-EF (VS) ≤ 0 H1: AUTO-EF (VF) - AUTO-EF (VS)> 0; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline in the Score of the Meta-memory in Adulthood Questionnaire - Portuguese Reduced Version
Description: The short version of Meta-memory in Adulthood Questionnaire is composed of 39 multiple-choice statements that are answered in a five-point likert scale, evaluating seven factors of meta-memory (strategy, task, capacity, change, anxiety, achievement and locus).
  Secondary Outcome Measures will evaluate the change from baseline of seven factors of meta-memory. The variation of the total sum obtained by means of the MIA questionnaire will be compared between all the visits in which the questionnaire was applied, ie, visit of selection (VS), visit 2 (V2) and final visit (VF).
Time Frame: 12 weeks after the start of the treatment (Baseline)
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in Stroop Test Victoria Version
Description: Change from Baseline in Stroop Test Victoria version
Time Frame: 12 weeks after the start of the treatment
Reporting Status: Not Posted

4. Secondary Outcome: The Overall Assessment of the Effectiveness of the Treatment by the Participant
Description: The overall assessment of the effectiveness of the treatment by the participant, through multiple-choice statements in a five-point likert scale
  1. My memory worsened in relation to the beginning of this treatment.
  2. There has been no improvement in my memory, which remains the same as when I started this treatment.
  3. My memory improved a little compared to how it was before the beginning treatment.
  4. My memory improved a lot compared to how it was before the beginning of this treatment.
  5. My memory returned to normal, that is, it returned to being as before the menopause.
Time Frame: 12 weeks after the start of the treatment
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Rate of Discontinuation of Treatment Due to Adverse Events.
Description: Rate of discontinuation of treatment due to adverse events.
Time Frame: 12 weeks after the start of the treatment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in Vital Signs (Blood Pressure) at the End of Treatment Compared to Baseline
Description: Changes in vital signs (blood pressure) at the end of treatment compared to baseline
  The blood pressure will be analyzed by the variation of the values measured at each visit in relation to the baseline value (VR), which will be summarized by means of descriptive statistics according to the treatment group.
Time Frame: 12 weeks after the start of the treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Changes in Vital Signs (Heart Rate) at the End of Treatment Compared to Baseline
Description: Changes in vital signs (heart rate) at the end of treatment compared to baseline
  The heart rate will be analyzed by the variation of the values measured at each visit in relation to the baseline value (VR), which will be summarized by means of descriptive statistics according to the treatment group.
Time Frame: 12 weeks after the start of the treatment
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Changes in Vital Signs (Respiratory Rate) at the End of Treatment Compared to Baseline
Description: Changes in vital signs (respiratory rate) at the end of treatment compared to baseline
  The respiratory rate will be analyzed by the variation of the values measured at each visit in relation to the baseline value (VR), which will be summarized by means of descriptive statistics according to the treatment group.
Time Frame: 12 weeks after the start of the treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Cogmax®
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 47/80
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cogmax® (N=80)
Gingivitis, Nasopharyngitis and Respiratory tract infection (Infections and infestations) | 2 (3)
Vascular disorders (Vascular disorders) | 25 (26)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 21 (37)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 18 (29)
Endocrine disorders (Endocrine disorders) | 8 (8)
Gastrointestinal disorders (Gastrointestinal disorders) | 8 (9)
Immune system disorders (Immune system disorders) | 5 (5)
Nervous system disorders (Nervous system disorders) | 3 (4)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (2)
Hepatobiliary disorders (Hepatobiliary disorders) | 2 (2)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (1)
Social circumstances (Social circumstances) | 1 (1)
Cardiac disorders (Cardiac disorders) | 1 (2)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 1 (1)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT03835325/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT03835325/SAP_001.pdf